CLINICAL TRIAL: NCT06331390
Title: Randomized Controlled Trial of Niacinamide Cosmetic Product Efficacy in Model of Irritant Contact Dermatitis
Brief Title: Assessment of Niacinamide Cosmetic Product Efficacy in Model of Irritant Contact Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Dario Leskur, assistant professor, University of Split, School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2181-198-03-04-24-0008
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervenition (Experimental): immortela cosmetic product
  Interventions: Other: niacinamide cosmetic product
- placebo (Placebo Comparator): nothing
  Interventions: Other: placebo

INTERVENTIONS:
Other: niacinamide cosmetic product — immortella skincare product
  Arms: intervenition
Other: placebo — nothing
  Arms: placebo

SUMMARY:
Testing the effectiveness and safety of cosmetics with niacinamide in irritant contact dermatitis: A Randomised, Controlled Trial will be conducted at USSM. Healthy volunteers will be included (at least 25) and test sites are forearms. Sodium lauryl sulphate will be used to induce contact dermatitis and participants will be measured for 7 days

DETAILED DESCRIPTION:
The efficacy of niacinamide cosmetic product on contact dermatitis will be evaluated using Courage Khazaka device and probes for hydration, redness and transepidermal water loss

ELIGIBILITY:
Inclusion Criteria:

* young, healthy volunteers who gave written informed consent

Exclusion Criteria:

* skin disease, skin damage on measurement sites, use of corticosteroids and immunomodulators a month prior to the inclusion and during the trial, non-adherence to the trial protocol, exposure to artificial UV radiation, pregnancy and lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
tewameter | day 1- day 7
  measurement of transepidermal water loss on skin, objective and non invasive

CONTACTS AND LOCATIONS:
Overall Officials: JOSIPA BUKIĆ, Principal Investigator — USSM
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided